CLINICAL TRIAL: NCT02865681
Title: Protocol to Minimize Injections and Blood Draws for Women Undergoing Controlled Ovarian Hyperstimulation for in Vitro Fertilization
Brief Title: Protocol to Minimize Injections and Blood Draws for Women Undergoing in Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Hope Fertility Center (Other)
Responsible Party: Principal Investigator, Zaher Merhi, M.D., Assistant Professor, New Hope Fertility Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JZ08-15
Record Dates: First submitted 2016-07-14; First posted 2016-08-12 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Infertility
Keywords: Infertility; Gonadotropins; Menopur; Ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — Menotropins; Gonadotropins; Nafarelin; Gonadotropin-Releasing Hormone; Clomiphene; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Conventional IVF (Active Comparator): Conventional ovarian stimulation consist of ovarian stimulation with daily gonadotropins injections daily starting in the early follicular phase (cycle day 3). The final maturation of oocytes will be induced with the standard hCG trigger when at least two follicles reached 18 mm or greater. Oocyte retrieval will be performed by either local or general anesthesia depending on the ovarian response, i.e., the number of mature follicles. Retrieved oocytes will be fertilized by IVF/ICSI and subsequently cultured until the blastocyst stage. All blastocysts will be vitrified. A single thawed blastocyst will be transferred in a subsequent natural or artificially prepared cycle.
  Interventions: Drug: Menopur; Drug: Synarel; Drug: HCG trigger; Drug: Clomiphene citrate; Drug: Letrozole
- IVF protocol using nasal gonadotropins (Experimental): Instead of injectable gonadotropins, nasal human menopausal gonadotropins (hMG; menopur) and oral clomiphene citrate and/or oral letrozole starting in the early follicular phase (cycle day 3). When at least two follicles reached 18 mm or greater, Synarel (Nafarelin) will be used instead of the injectable HCG trigger. Oocyte retrieval will be performed by either local or general anesthesia depending on the ovarian response, i.e., the number of mature follicles. Retrieved oocytes will be fertilized by IVF/ICSI and subsequently cultured until the blastocyst stage. All blastocysts will be vitrified. A single thawed blastocyst will be transferred in a subsequent natural or artificially prepared cycle.
  Interventions: Drug: Menopur; Drug: Synarel; Drug: Clomiphene citrate; Drug: Letrozole

INTERVENTIONS:
Drug: Menopur — Nasal versus injectable
  Other Names: gonadotropin
Drug: Synarel — nasal
  Other Names: GnRH agonist
Drug: HCG trigger — injectable
  Other Names: HCG
  Arms: Conventional IVF
Drug: Clomiphene citrate — oral
  Other Names: Clomid
Drug: Letrozole — Oral
  Other Names: Femara

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of nasal gonadotropins (Menopur) in women undergoing IVF. The purpose of this study is also to report and monitor any and all side effects of the nasal Menopur.

DETAILED DESCRIPTION:
Gonadotropins are used during fertility treatments such as intrauterine insemination (IUI) or in vitro fertilization (IVF). These fertility medications are given by injection that contain follicle-stimulating hormone (FSH) alone or combined with luteinizing hormone (LH). During a regularly occurring menstrual cycle, both FSH and LH are produced by the pituitary gland in the brain to naturally stimulate the ovaries to make a single egg each month. When FSH and/or LH are given as an injection as fertility treatment, they work directly on the ovaries to make multiple follicles which are cysts containing the eggs.

Injections of gonadotropins are started early (usually on the third day) in the menstrual cycle to cause multiple eggs to grow to a mature size. Close monitoring of patients with ultrasound and blood are usually needed for monitoring. The ultrasound measures the size of the ovarian follicles. Blood is usually drawn every other day or daily (for a total of 12 days on average) for measurement of Estradiol (E2), progesterone (P4), and luteinizing hormone (LH). The measurement of E2, P4 and LH is intended to quantify the response of the ovaries to the daily injectable gonadotropins. When the follicles grow to a large size (usually 18 mm), human chorionic gonadotropin (hCG), another injectable medication, is then used to trigger the maturity of the eggs before performing egg retrieval during an IVF cycle.

Instead of injectable gonadotropins, this study uses nasal gonadotropins (Menopur) in order to evaluate its safety and efficacy of in women undergoing IVF.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-45. The participant should be a woman of reproductive age, i.e., premenopausal who is healthy.
2. Body mass index: 19-35 kg/m2
3. Diagnosis of infertility: inability to conceive with unprotected intercourse after 1 year for women aged < 35 and after 6 months for women aged > 35.
4. Pap smear within 1 year should be normal.
5. Endometrial cavity will be evaluated and should be normal using hysteroscopy or saline ultrasound
6. Fallopian tubes will be assessed by hysterosalpingogram in women who have normal ovarian reserve, regular menstrual cycles with a partner who has normal semen analysis. Unless there is a clear diagnosis of a reason for infertility, such as poor sperm, poor ovarian reserve, fallopian tube patency will not be performed because it would not change the treatment.
7. Semen analysis will be performed on every male partner to ensure that there are sperm to be used for IVF/ICSI.
8. All assessment will be performed at baseline and before initiation of any treatment.
9. The investigators will obtain at screening Pap smear, hysteroscopy or saline ultrasound, hysterosalpingography, and semen analysis if they have not been done within one year of baseline.

Exclusion Criteria:

1. Any medical condition that interferes with the health of the participant such as uncontrolled diabetes, uncontrolled hypertension, cardiac disease, or renal disease.
2. Any type of malignancy.
3. Mental problems that could interfere with the patient's ability to conceive and take care of her baby.
4. Abnormal endometrial cavity that could interfere with implantation and/or carrying the pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Serum estradiol level | 1 year
  serum estradiol level in pg/mL as representative of ovarian response
Ovarian follicular size | 1 year
  Pelvic ultrasound to measure the size of each ovarian follicle as representative of ovarian response

SECONDARY OUTCOMES:
Adverse Events That Are Related to Nasal Menopur Treatment | 1 year
  whether there are any side effects

CONTACTS AND LOCATIONS:
Locations (1):
- New Hope Fertility Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
will share the data upon request

REFERENCES:
- [Result] Zhang J, Merhi Z. Safety data for the use of nasal human menopausal gonadotropins: a potential novel approach for fertility treatment. JBRA Assist Reprod. 2019 Apr 30;23(2):169-171. doi: 10.5935/1518-0557.20180078. PMID 30500132